CLINICAL TRIAL: NCT01968720
Title: A Phase 2 Pilot Study to Assess the Safety and Efficacy of CAT-2003 in Patients With Severe Hypertriglyceridemia
Brief Title: Pilot Study To Assess CAT-2003 in Patients With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CAT-2003-202
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Hyperlipidemias; Hypertriglyceridemia; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Hyperlipidemias; Hypertriglyceridemia; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAT-2003 or Placebo (Experimental): All patients will receive placebo for a 14 day treatment period and CAT-2003 for a 28 day treatment period.
  Interventions: Drug: CAT-2003; Drug: Placebo

INTERVENTIONS:
Drug: CAT-2003
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of multiple doses of CAT-2003 in patients with severe hypertriglyceridemia either naive or refractory to current therapy. The study will evaluate effects of CAT-2003 on fasting and postprandial total triglycerides and chylomicron triglyceride levels in patients with severe hypertriglyceridemia.

This is a single-blind study. All patients will receive placebo for a 14 day treatment period and CAT-2003 for a 28 day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 74 years at Screening
* Severe Hypertriglyceridemia (TG ≥ 500 mg/dL). If on lipid lowering therapy including statins, fibrates, and/or omega-3 fatty acids, stable dose for at least 4 weeks prior to Screening
* Body mass index (BMI) ≤ 45 kg/m2

Exclusion Criteria:

* History of any major cardiovascular event within 6 months of Screening
* Type I diabetes mellitus or use of insulin
* History of pancreatitis

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in fasting triglycerides in patients with severe hypertriglyceridemia | 4 weeks

SECONDARY OUTCOMES:
Frequency of adverse events | 4 weeks
  Safety will be assessed for all enrolled patients from the time the patient signs the informed consent through post-treatment follow-up.
  Safety parameters include physical exam, vital signs, clinical laboratory tests, ECGs and concomitant medications.
Absolute and percent change from baseline on postprandial total and chylomicron triglyceride levels | 4 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Miami, Florida
  - Indianapolis, Indiana
  - Auburn, Maine
  - Cincinnati, Ohio